CLINICAL TRIAL: NCT00745160
Title: Survey and Blood Sample Collection for Patients With Lung Cancer Who Never Smoked Cigarettes
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Vincent Miller, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 08-104
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: Questionaires
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample for DNA analysis

GROUPS / COHORTS (1):
- 1: Never-smokers with lung cancer
  Interventions: Other: blood sample and questionnaire

INTERVENTIONS:
Other: blood sample and questionnaire — After giving informed consent, all patients will be asked to complete questionnaire and will be asked to provide a blood sample for DNA analysis. The questionnaire will consist of a detailed smoking questionnaire, based on the most recent Centers for Disease Control and Prevention (CDC) Behavioral Risk Factor Surveillance System Survey Questionnaire.

SUMMARY:
The purpose of this study is to determine if collecting information and blood from a group of people who never smoked but who have lung cancer, is possible across the US. The investigators will collect information on each patient's diagnosis and treatments. If the collection is successful, blood samples will be used to try to identify new genes (which are the basic elements of heredity, passed from parents to their offspring), which may explain and predict why certain patients develop lung cancer without having smoked tobacco.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* histologically and/or cytologically proven diagnosis of non-small cell lung cancer
* never smoker, defined as having smoked less than 100 cigarettes over one's life-time
* completed survey and inclusion form
* signed informed consent

Exclusion Criteria:

* previous history of cancer (other than lung cancer)
* living outside the United States
* patients who cannot read English (as website and questionnaires will only be written in English)
* unable to understand the protocol or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Never-smokers with lung cancer
  Internet recruitment The study will be advertised through a specifically designed website linked to the MSKCC Lung Cancer webpage. The website will be designed after approval of the study. The website will be accordingly reviewed by the IRB. We plan to advertise this study by word-of mouth at scientific meetings and on patient associations' websites and/or bulletins, with permission. The website will post a description of the study and an invitation to participate.
  Interested patients will be given an email or mail address and/or phone number 866-854-4652 to contact MSKCC investigators about the study.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of an internet-based protocol to collect clinical information and biological specimens from 2,000 never smokers with lung cancer. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Miller, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York